CLINICAL TRIAL: NCT05818917
Title: A Phase 1, Multi-Center, Open-Label Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Preliminary Evidence of Antitumor Activity of FHND5071 as a Single Agent in Adult Patients With Advanced Solid Tumors
Brief Title: A Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Preliminary Evidence of Antitumor Activity of FHND5071 as a Single Agent in Adult Patients With Advanced Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Jiangsu Chia Tai Fenghai Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: FHND5071-I-01
Record Dates: First submitted 2023-03-29; First posted 2023-04-19 (Actual); Last update posted 2023-04-19 (Actual); Status verified 2023-04

CONDITIONS: Advanced Solid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- 40mg (Experimental): FHND5071, 40mg, tablet, orally, once daily
  Interventions: Drug: FHND5071
- 80mg (Experimental): FHND5071,80mg, tablet, orally, once daily
  Interventions: Drug: FHND5071
- 160mg (Experimental): FHND5071, 160mg, tablet, orally, once daily
  Interventions: Drug: FHND5071
- 240mg (Experimental): FHND5071, 240mg, tablet, orally, once daily
  Interventions: Drug: FHND5071
- 320mg (Experimental): FHND5071, 320mg, tablet, orally, once daily
  Interventions: Drug: FHND5071
- 400mg (Experimental): FHND5071, 400mg, tablet, orally, once daily
  Interventions: Drug: FHND5071

INTERVENTIONS:
Drug: FHND5071 — The proposed starting dose is 40 mg FHND5071 once daily (QD) orally (PO). For the purposes of this study treatment cycles will be 28 days or 4 weeks.
  FHND5071 will be administered orally in the morning following a fast of approximately 10 hours before dosing on PK collection days. Subjects will continue to fast for approximately 4 hours after the administration of FHND5071. On non-PK days the subjects will fast approximately 2 hours before FHND5071 and continue to fast for approximately 2 hours afterwards.
  Other dosing regimens may be considered based on the analysis of emerging PK, progressive disease, and/or safety data.

SUMMARY:
This is a Phase 1, first-in-human, open-label dose-escalation study to determine the MTD and/or recommended Phase 2 dose (RP2D) and assess the DLT of FHND5071. The safety, tolerability, and PK of FHND5071 will be assessed in adult patients with advanced solid tumors.

The total number of evaluable subjects in the study will depend upon the number of dose-escalations necessary. It is estimated that approximately 24 evaluable subjects will be enrolled in the dose-escalation part of this study. This multicenter study will be conducted in the United States.

Dose-escalation of FHND5071 will follow two sequential parts:

1. a modified accelerated titration design in single subject cohorts with a starting dose level of 40 mg, where the FHND5071 dose would be doubled in each dose cohort until the subject in a current cohort experience a Grade ≥2 adverse event that is at least possibly related to FHND5071 in the opinion of the Investigator and the Medical Monitor;
2. a modified 3+3 escalation design in cohort of 3-6 subjects, where the FHND5071 dose would be escalated in ≤100% increments determined by the Safety Review Committee (SRC) until 2 of 3 or 2 of 6 subjects experience a DLT. In both parts of dose escalation, FHND5071 will be administered orally once daily (QD) in 28-day treatment cycles.

Escalation cohorts may explore alternative doses or different schedules, if deemed appropriate by the Safety Review Committee.

ELIGIBILITY:
Inclusion Criteria:

Only the subjects who meet all of the following inclusion criteria are eligible for entry into this study:

1. The subjects agree and have the ability to comply with the study and follow-up procedures. Before any examination and study, the subjects or their legal guardians shall sign and date a written informed consent;
2. Age ≥ 18 years old, male or female;
3. The Eastern Cooperative Oncology Group Performance Status (ECOG PS) score is 0~1;
4. The expected survival period is not less than 12 weeks;
5. Subjects have at least one evaluable lesion according to RECIST V1.1. Tumor lesions that have progressed after being irradiated ≥4 weeks before the start of treatment can be used as target lesions in the absence of non-irradiated evaluable lesions;
6. Subjects with advanced solid tumors confirmed by histology or cytology, for whom the standard treatment has failed, or there is no standard treatment regime, or the standard treatment is not applicable at the current stage;
7. Subjects must have adequate organ functions, as defined below:

   Liver function:

   •Serum aspartate aminotransferase (AST), serum alanine aminotransferase (ALT) ≤ 2.5 times the upper limit of normal (ULN); total serum bilirubin (TBIL) ≤ 1.5 times ULN (for subjects with Gilbert syndrome, serum bilirubin ≤ 3.0 × ULN).

   Bone marrow function (no blood transfusion or hematopoietic stimulating factor therapy within 10 days prior to testing):
   * Absolute neutrophil count (ANC) ≥1.5×109/L;
   * Platelet (PLT) ≥100×109/L;
   * Hemoglobin (Hb) ≥9g/dL;
   * Lymphocyte count ≥0.5×109/L.

   Kidney function:

   •Serum creatinine ≤1.5 mg/dL, or estimated glomerular filtration rate ≥60 mL/min/1.73m2 using the Chronic Kidney Disease Epidemiology Partnership (CKD-EPI) formula;

   Coagulation:

   If the subject does not take anticoagulants, INR < 1.5. If the subject is taking anticoagulants, INR < 3.
8. For fertile women, the serum pregnancy test must be negative prior to the enrollment into the study. Infertile women who have had natural (instinctive) menopause for at least 12 consecutive months prior to screening, with appropriate clinical manifestation (e.g. appropriate age, history of vasomotor symptoms), or have undergone bilateral oophorectomy, hysterectomy or bilateral tubal ligation more than 6 weeks prior to screening;
9. Male or female subjects: Male subjects (whose partner is a fertile female) and fertile female subjects must use two acceptable methods of contraception, including one barrier method, throughout the study period until 3 months after the last dose. Male subjects must also avoid donating sperm while participating in the study;
10. Subjects must be able to swallow and absorb oral medication.

Exclusion Criteria:

Subjects who meet any of the following will not be able to enter this study:

1. Previous (≤3 years) or current existence of cancer histologically determined to be different from the study tumors, except for cervical carcinoma in situ, superficial non-invasive bladder tumor, or cured stage I non-melanoma skin cancer;
2. Subjects carrying known major mutational driver genes other than RET gene, such as: EGFR, ALK, ROS1, etc.;
3. Known severe allergy to the study drug or excipient (microcrystalline cellulose);
4. Severe autoimmune diseases (including immune-related AEs from previous immuno-oncology therapy) or autoimmune diseases requiring chronic systemic corticosteroid therapy with immunosuppressive doses (prednisone >10 mg/day or equivalent);
5. Known malignant central nervous system diseases, except for neurologically stable and treated brain metastases, which are defined as brain metastases that have been treated with surgery, surgery plus radiotherapy, or radiotherapy alone, with no signs of progression or hemorrhage within 14 days after treatment and all systemic corticosteroids discontinued within 14 days prior to the treatment.
6. Medical history (within 6 months before treatment initiation) or evidence of pericarditis (of any grade) or pericardial effusion (≥ Grade 2);
7. Medical history (within 6 months prior to initiation of therapy) or evidence of interstitial lung disease, radiation pneumonitis or idiopathic pulmonary fibrosis requiring steroid therapy, pleural or pericardial effusion requiring intervention such as drainage.
8. Medical history (within 4 weeks after initiation of therapy) or evidence of active infection (≥ Grade 2);
9. Medical history of positive serostatus for human immunodeficiency virus (HIV), hepatitis B virus (HBV), or hepatitis C virus (HCV) at any time before treatment:

   * Positive anti-HIV-1 or anti-HIV-2 antibodies,
   * or positive HBsAg
   * or positive anti-HCV antibody or quantifiable HCV-RNA.
   * For subjects with no previous result report, whether to conduct testing of serostatus during the screening period will be at the discretion of the investigator;
10. Medical history (≤6 months before treatment) or evidence of any serious and/or uncontrolled medical condition or circumstances that the investigator and sponsor believe may affect the subject's participation in the study, for example:

    * Non-malignant disease that is not under control or the existing disease control of which could be jeopardized by the treatment in this study;
    * Malignant decompensated liver disease;
    * Severe gastrointestinal abnormalities or chronic diseases that affect absorption or intravenous nutritional needs, including inability to swallow formula products, delayed gastric emptying, chronic diarrhea associated with intestinal malabsorption, ulcerative colitis, or Crohn's disease requiring any dose level of steroids, refractory nausea and vomiting, and/or prior surgery.
11. With medical history (≤6 months before treatment initiation) or evidence of any of the following: acute myocardial infarction, unstable angina, coronary artery bypass grafting, cerebrovascular accident, or transient cerebral ischemic attack;
12. Subjects with impaired cardiac function or clinically significant cardiac diseases, including any of the following; congenital long QT syndrome;

    * Severe ventricular or supraventricular arrhythmia (in the absence of other cardiac abnormalities, atrial fibrillation patients with sinus arrhythmia or slow ventricular rate are eligible);
    * LVEF<50% evaluated by ECHO or MUGA;
    * Resting bradycardia (<50 beats per min) is determined by the mean of 3 heart rate values from three qualified ECG screenings;
    * Other serious heart diseases, such as congestive heart failure of Class III-IV according to New York Heart Association (NYHA);
13. Subjects with a QT interval >470 ms corrected by the Fridericia formula (determined by the mean of 3 QTcF values from three qualified ECG screenings) during the screening phase;
14. Medical history (≤6 months before treatment) or evidence of concomitant diseases that may prolong the QT interval according to the judgment of investigators and medical monitors;
15. Medical history (≤6 months before treatment) or evidence of severe inflammatory or vascular ocular diseases (e.g., retinal vein occlusion);
16. Subjects with unhealed toxicity higher than Grade 1 before treatment, except for those with hair loss (alopecia), Grade 2 neuropathy (if permitted by the investigator) or hemoglobin of 9-10 g/dL;
17. Medical history (≤6 months before treatment) or evidence of malignant biliary obstruction, except for those with normal biliary stent function:
18. Pregnant or breastfeeding women;
19. History of bone marrow transplant or solid organ transplant;
20. Use of systemic anticancer drugs (except for the antiandrogen therapy treating prostate cancer) or study drugs within 28 days prior to the first dose of FHND5071;
21. Medical history of radiation therapy within 28 days prior to the first dose of FHND5071, or radiation therapy possibly required at any time until 30 days after the last dose of FHND5071, except for palliative radiation therapy limited to non-targeted lesions;
22. Medical history (within 28 days after the treatment starts) or evidence of major surgery or trauma, or potentially required surgery during treatment (the severity will be determined by the investigator in consultation with the medical monitor) ;
23. Medical history of transfusion of whole blood, red blood cells or platelets within 2 weeks before the start of treatment;
24. Patients using erythropoietin or granulocyte colony-stimulating factor (G-CSF), filgrastine or filgrastine for less than or equal to 2 weeks before treatment;
25. Medical history of medication known to have risk of inducing torsades de pointes (arrhythmia due to drug-induced QTc prolongation) within 2 weeks before treatment until EOT follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-07-07 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Reporting One or More Treatment-Emergent Adverse Events and Serious Adverse Events | Baseline to 28 days after first dose of FHND5071 administration
  An Adverse Event is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (eg, a clinically significant abnormal laboratory finding), symptom, or disease temporally associated with the use of a drug, whether or not it is considered related to the drug. A treatment-emergent adverse event (TEAE) is defined as an adverse event with an onset that occurs after receiving study drug. A Serious Adverse Event (SAE) was any experience that suggests a significant hazard, contraindication, side effect or precaution that: results in death, is life-threatening, required in-patient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect or is medically significant.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Shanghai Chest Hospital, Shanghai
  - Tianjin People's Hospital, Tianjin

IPD SHARING:
Plan to Share IPD: No